CLINICAL TRIAL: NCT05219266
Title: Managed Access Programs for PKC412, Midostaurin
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CPKC412A2407I
Record Dates: First submitted 2021-10-05; First posted 2022-02-02 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: FMS-Like Tyrosine Kinase 3 (FLT3)-Mutated Acute Myeloid Leukemia; Acute Myeloid Leukemia; Aggressive Systemic Mastocytosis; Mast Cell Leukemia; Systemic Mastocytosis With an Associated Hematologic Neoplasm
Keywords: FLT3-mutated AML; AML; Aggressive systemic mastocytosis; Mast cell leukemia; Systemic mastocytosis with an associated hematologic neoplasm; MAP; Manage access program; PKC412; Midostaurin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Mastocytosis, Systemic; Leukemia, Mast-Cell | interventions — midostaurin

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: midostaurin — Patients receive midostaurin
  Other Names: PKC412

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to PKC4, Midostaurin.

DETAILED DESCRIPTION:
* CPKC412A2001X - No longer available- An open-labeled, multi-center, Expanded Treatment Protocol (ETP) of midostaurin (PKC412) in patients 18 years of age or older with newly-diagnosed FLT3-mutated acute myeloid leukemia (AML) who are eligible for standard induction and consolidation chemotherapy
* CPKC412AUS56X - No longer available - An open-label, multi-center, Expanded Treatment Protocol of Midostaurin (PKC412) in adult patients with newly diagnosed Fms-like tyrosine kinase receptor (FLT3) mutated Acute Myeloid Leukemia (AML) who are eligible for standard induction and consolidation chemotherapy.
* CPKC412A2407I - No longer available- Managed Access Program (MAP) Cohort Treatment Plan CPKC412A2407I to provide access to midostaurin (PKC412) for patients 18 years of age and older with newly-diagnosed FLT3-mutated AML and eligible for induction and consolidation chemotherapy
* CPKC412D2001M - No longer available- Managed Access Program (MAP) to provide access to Midostaurin (PKC412), for an individual patient with aggressive systemic mastocytosis (ASM), mast cell leukemia (MCL) or mast cell sarcoma (MCS)

ELIGIBILITY:
Inclusion Criteria:

* An independent request should be received from a licensed physician (in some instances from Health Authorities, Institutions or Governments).
* The patient has a serious or life-threatening disease or condition and no comparable or satisfactory alternative therapy is available for diagnosis, monitoring or treatment; patient is not medically eligible for available treatment alternatives or has exhausted all available treatment options.
* The patient is not eligible or able to enroll in a Novartis clinical trial or continue participation in a Novartis clinical trial.
* There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
* The patient must meet any other medical criteria established by the medical experts responsible for the product or by the Health Authority in a country (as applicable).
* Provision of the product will not interfere with the initiation, conduct or completion of a Novartis clinical trial or overall development program.
* Managed access provision is allowed per local laws/regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult